CLINICAL TRIAL: NCT01779856
Title: Monitoring in Dialysis
Brief Title: Monitoring in Dialysis -- a Prospective, Multi-center, Single-arm, Non-randomized, Observational Study in Patients Who Are Undergoing Hemodialysis.
Acronym: MiD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Corporate Technologies and New Ventures (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: G120171
Record Dates: First submitted 2013-01-22; First posted 2013-01-30 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease, Hemodialysis, Arrhythmia, Reveal ICM
MeSH Terms: conditions — Kidney Failure, Chronic; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- REVEAL Insertable Cardiac Monitor (ICM) (Other): Monitoring of cardiac arrhythmic events and the relationship between such events and the characteristics.
  Interventions: Device: REVEAL Insertable Cardiac Monitor (ICM)

INTERVENTIONS:
Device: REVEAL Insertable Cardiac Monitor (ICM)
  Other Names: Reveal ICM

SUMMARY:
The primary objective of this study is to estimate the proportion of hemodialysis patients experiencing clinically significant cardiac arrhythmias over a 6-month period using continuous cardiac monitoring with an implanted Medtronic Reveal Insertable Cardiac Monitor (ICM) device.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older and is willing to be implanted with the Reveal ICM
* Currently on hemodialysis at least three times per week OR has an estimated glomerular filtration rate (eGFR) of < 15 mL/min/1.73m^2 and is expected to begin hemodialysis within 2 months.
* Subject is willing and able to comply with the protocol

Exclusion Criteria:

* Currently enrolled in an interventional study that may interfere with the Monitoring in Dialysis protocol
* Not suitable for Reveal ICM implantation
* Has an existing hemodialysis catheter that may interfere with the Reveal ICM implantation site
* Has a recent infection
* Is currently on hemodialysis with a hemoglobin < 10 g/dL
* Has end-stage liver failure or has had thoracic surgery within the past 6 months
* Has an existing pacemaker, implantable cardioverter-defibrillator (ICD) or cardiac resynchronization device
* Is scheduled for renal transplantation or will likely be transplanted within 6 months
* Is currently on home hemodialysis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Augusta, Georgia
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Chattanooga, Tennessee
  - Houston, Texas
- India (4):
  - Chennai
  - Gūrgaon
  - Hyderabad
  - New Delhi

REFERENCES:
- [Derived] Soomro QH, Bansal N, Winkelmayer WC, Koplan BA, Costea AI, Roy-Chaudhury P, Tumlin JA, Kher V, Williamson DE, Pokhariyal S, McClure CK, Charytan DM; MiD Investigators. Association of Bradycardia and Asystole Episodes with Dialytic Parameters: An Analysis of the Monitoring in Dialysis (MiD) Study. Kidney360. 2022 Oct 11;3(11):1871-1880. doi: 10.34067/KID.0003142022. eCollection 2022 Nov 24. PMID 36514397
- [Derived] Tumlin JA, Roy-Chaudhury P, Koplan BA, Costea AI, Kher V, Williamson D, Pokhariyal S, Charytan DM; MiD investigators and Committees. Relationship between dialytic parameters and reviewer confirmed arrhythmias in hemodialysis patients in the monitoring in dialysis study. BMC Nephrol. 2019 Mar 5;20(1):80. doi: 10.1186/s12882-019-1212-6. PMID 30836948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects on dialysis 3 times per week
Groups:
- REVEAL Insertable Cardiac Monitor (ICM): Patients implanted with Medtronic Reveal XT or LINQ Device
Period: Overall Study
Arm/Group | REVEAL Insertable Cardiac Monitor (ICM)
Started | 81
Completed | 57
Not Completed | 24
Not completed — Withdrawal by Subject | 15
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Inclusion/Exclusion Not Met | 2
Not completed — Delays in scheduling implant | 1
Not completed — Subject ineligible for Implant | 2

BASELINE CHARACTERISTICS:
Population: Number of subjects who were eligible for implant after consent
Groups:
- REVEAL Insertable Cardiac Monitor (ICM): Monitoring of cardiac arrhythmic events and the relationship between such events and the characteristics.
  REVEAL Insertable Cardiac Monitor (ICM)
Arm/Group | REVEAL Insertable Cardiac Monitor (ICM)
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 28
  Black or African American | 39
  White or Caucasian | 7
Region of Enrollment [Number; unit: participants]
  United States | 47
  India | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Cardiac Arrhythmias Using Continuous Cardiac Monitoring Over a 6-month Period With an Implanted Medtronic Reveal ICM Device
Description: Events defined as clinically significant for the objective include: episodes of ventricular tachycardia (VT) greater than or equal to 130 beats per minute (BPM), episodes of bradycardia indicated by a recorded heart rate less than or equal to 40 BPM, instances of asystole lasting at least three seconds, or any symptomatic event, indicated by patient use of the Reveal ICM Patient Assistant, where review of the stored ECG shows an arrhythmia considered clinically significant in the judgement of the study site cardiologist.
Time Frame: 6 months of dialysis data following Reveal ICM implant
Population: 81 subjects were enrolled in the study; however, only 66 subjects were implanted with the device. This accounts for the difference in analyzed numbers.
Measure: Number; unit: participants
Arm/Group | REVEAL Insertable Cardiac Monitor (ICM)
Number analyzed (Participants) | 66
participants
  All CSA | 44
  CSA Subtype (VT) | 1
  CSA Subtype (Bradycardia) | 13
  CSA Subtype (Asystole) | 6
  CSA Subtype (Patient Marked Events) | 38

2. Secondary Outcome: Collect the Number of Device and Procedure Related Adverse Events (AEs).
Description: All procedure and device-related AEs will be recorded as they occur, and will be categorized according to seriousness, intensity, and relatedness to the device, device components, or implant procedure.
Time Frame: 6 months of dialysis data following Reveal ICM implant
Measure: Number; unit: Events
Groups:
- Adverse Events: Study Subjects with Adverse Events
Arm/Group | Adverse Events
Number analyzed (Participants) | 81
Events
  Procedure Releated AEs | 3
  Device Related AEs | 2
  Not Related | 50
  Unknown | 2

3. Secondary Outcome: Nature and Time of Health-related Events and Treatment Associated With ESRD and Other Conditions Occurring in the Implanted Patients
Description: Health-related events were recorded as they occurred. All health-related events were tabulated and summarized by type, time of occurrence (first 6 months and All Available Time (up to 2 years) and number of subjects affected.
Time Frame: up to 6 months and through study completion
Population: Health-related events were recorded as they occurred. All health-related events were tabulated and summarized by type, time of occurrence, number of occurrences, and number of subjects affected. Summary statistics include events counts.
Measure: Number; unit: number of events reported by
Groups:
- First 6 Months of Follow-up: Number of health care utilizations, by category, that occurred within the first 6 months of follow-up
- All Available Time (up to 2 Years): Number of health care utilizations, by category, that occurred within the course of the study.
Arm/Group | First 6 Months of Follow-up | All Available Time (up to 2 Years)
Number analyzed (Participants) | 81 | 81
number of events reported by
  Inpatient : number of events reports | 33 | 44
  Out-Patient : number of events reports | 14 | 15
  Emergency Department : number of events reports | 35 | 42
  Urgent Care : number of events reports | 57 | 73

4. Secondary Outcome: Rate of Arrhythmias by Intradialytic Potassium Change and Volume Removed
Description: The atrial arrhythmic events, ventricular arrhythmic events, and AF burden were tabulated and reported. Atrial arrhythmic episodes were distributed temporally over the inter- and intradialytic periods using the negative binomial mixed effect regression model as described above in the primary objective analysis.
Time Frame: 6 Month Follow-up
Population: Reviewer confirmed arrhythmia rate normalized per hour
Measure: Number; unit: arrhythmic events
Groups:
- Volume Removed 2.3; Volume Removed 3.3; Volume Removed 4.3: (L) volume removed during dialysis
Arm/Group | Volume Removed 2.3 | Volume Removed 3.3 | Volume Removed 4.3
Number analyzed (Participants) | 66 | 66 | 66
arrhythmic events
  0 Potassium Change | 0.013 | 0.02 | 0.007
  -1 Potassium Change | 0.014 | 0.015 | 0.016
  -2 Potassium Change | 0.015 | 0.023 | 0.03

5. Secondary Outcome: Collect and Quantify the Episodes of Arrhythmias
Description: The atrial arrhythmic events, ventricular arrhythmic events, and AF burden will be tabulated and reported.
Time Frame: 6 months of dialysis data following Reveal ICM implant
Measure: Number; unit: Arrhythmia Episodes
Arm/Group | REVEAL Insertable Cardiac Monitor (ICM)
Number analyzed (Participants) | 66
Arrhythmia Episodes
  Overall Reviewer Confirmed Arrhythmias | 64
  Atrial Fibrillation Arrhythmia > 6 min | 60
  Ventricular Arrhythmia | 51
  Bradycardia | 17
  Asystole | 7
  Sinus Tachycardia | 53
  Patient Marked | 38

6. Secondary Outcome: Assess Whether the Morphology of ECG Recordings Captured by the Reveal ICM Device Correlate With Serum Electrolyte Levels Measured Just Before and Just After Dialysis Sessions.
Description: The Reveal patient Assistant will be used to trigger memory storage of 7.5 minute ECG recordings in conjunction with serum electrolyte measurements taken before and after selected dialysis sessions. Measures of ECG morphology (e.g., QT interval, QT dispersion, QRS width, T-wave amplitude) will then be extracted from the recorded ECG data. The serum electrolyte data will also be included.
Time Frame: 6 months
Measure: Median (Full Range); unit: Correlation Coefficient
Groups:
- ECG Recording Captured by the Reveal ICM Device: Patients implanted with Medtronic Reveal XT or LINQ Device
Arm/Group | ECG Recording Captured by the Reveal ICM Device
Number analyzed (Participants) | 35
Correlation Coefficient
  R Value: R Wave Amplitude vs Potassium | -0.35 [-0.86 to 0.67]
  R Value: R Wave Amplitude vs Magnesium | -0.33 [-0.83 to 0.48]
  R Value: R Wave Amplitude vs. Phosphorus | -0.45 [-0.84 to 0.68]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 1 year.
Arm/Group | REVEAL Insertable Cardiac Monitor (ICM)
All-Cause Mortality (participants affected / at risk) | 3/81
Serious Adverse Events (participants affected / at risk) | 28/81
Other Adverse Events (participants affected / at risk) | 8/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REVEAL Insertable Cardiac Monitor (ICM) (N=81)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 3 (3)
Sinus arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Graft dysfunction (Injury, poisoning and procedural complications) | 2 (2)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 1 (1)
Renal transplant (Surgical and medical procedures) | 2 (2)
Accelerated hypertension (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Aortic dissection (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REVEAL Insertable Cardiac Monitor (ICM) (N=81)
Suture related complication (Surgical and medical procedures) | 1 (1)
Implant site pain (General disorders) | 2 (2)
Implant site haematoma (General disorders) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Impaired healing (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The intent of the project is to develop a foundation, which is scientifically based, to generate hypotheses resulting from data collected during theobservational study. Further research may be investigated based on the outcome of this small study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No